CLINICAL TRIAL: NCT05822778
Title: Safety and Efficacy Study of Formaderm (Hyaluronic Acid) for Facial Soft Tissue Augmentation
Brief Title: Formaderm (Hyaluronic Acid) for Facial Soft Tissue Augmentation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Maxigen Biotech Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Other
Other Study IDs: 2-102-05-113
Record Dates: First submitted 2023-03-16; First posted 2023-04-21 (Actual); Last update posted 2023-04-21 (Actual); Status verified 2023-04

CONDITIONS: Dermal Filler
Keywords: hyaluronic acid filler; nasolabial folds

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Formaderm(FD) group (Experimental): Formaderm was randomly administered either side of subjects' facial areas once. The injection volume was limited to 2c.c.
  Interventions: Device: Formaderm Dermal Filler Injection
- control group (Active Comparator): As a self-controlled study, "Q-MED" RESTYLANE would be administered on the other side after injected Formaderm. The injection volume was limited to 2c.c.
  Interventions: Device: "Q-MED" RESTYLANE

INTERVENTIONS:
Device: Formaderm Dermal Filler Injection — Dermal filler injection to facial areas
  Arms: Formaderm(FD) group
Device: "Q-MED" RESTYLANE — Dermal filler injection to facial areas
  Arms: control group

SUMMARY:
The goal of this clinical trial is to evaluate the safety and efficacy of Formaderm (hyaluronic acid) dermal filler injection for soft tissue augmentation. The main questions it aims to answer are:

* The differences of Wrinkle Severity Rating Scale (WSRS) after the injection.
* The differences of Global Aesthetic Improvement Scale (GAIS) after the injection.
* The subjective satisfaction of treatment.
* Safety Indicators of which incidences on the day of the injection or after the injection.

Participants will be self-controlled and randomized for same period

* received both trial product and control product at the same time.
* re-visited on week 2, 4, 12, 24, 36, and 52 after injection.

Researchers will compare if the test product is non-inferiority to Q-Med Restylane.

DETAILED DESCRIPTION:
The purpose of this study is to evaluate the safety and efficacy of Formaderm (hyaluronic acid) dermal filler injection for soft tissue augmentation. A single-centre, non-inferior, randomized, double-blind trial with a control group was conducted in this study. Every subject received the trial product and control product injections at the same time. It was planned to recruit 95 subjects with the 10% dropout rate. This clinical trial is accordance with the "Good Clinical Practice (GCP) issued by the Department of Health and ISO14155-1：2003 Clinical investigation of medical devices for human subjects - Part 1: General Requirements and carried out according to the trial proposal approved by the Tri-Service General Hospital Human Subjects Review Committee.

ELIGIBILITY:
Inclusion Criteria:

* Subjects are aged 30-65 years old of both sexes.
* Subjects who are willing to undergo WSRS therapy.
* The WSRS baseline measurement should be 3-4 points and the left and right side should be in symmetry.
* The facial skin is healthy, without any disease that possibly interferes with skin aging status assessment.
* The subject is willing to avoid undergoing other cosmetic treatment and surgery, including Botox injection.

Exclusion Criteria:

* Women subjects who are pregnant, breastfeeding, planning to become pregnant, and not willing to take contraception during the trial period.
* Those who are emotionally unstable or suffering from a mental disease.
* Those who have severe skin disease, inflammation, or related symptoms such as infections, psoriasis, herpes, and the like.
* Those who have undergone cosmetic treatment or surgery prior to the trial:
* Those who have undergone laser treatment or dermabrasion within the past 12 months.
* Those who have undergone chemical peels treatment within the last three months.
* Those who have undergone facial wrinkle augmentation surgery such as Botox injections within the past 12 months.
* Those with silicone in their body or material that cannot be absorbed by the body (permanent filling agent).
* Those who have undergone facial surgery or filing agent implants in the nasolabial fold area within the past 24 months.
* Those who have a scar or localized infection in the nasolabial fold area.
* Those with connective tissue diseases.
* Those with diabetes or systemic disease that cannot be controlled.
* Those suffering from human immunodeficiency syndrome.
* Those suffering from immunity related disorder or have had immune system degradation in the past.
* Those with a scar-prone constitution, prone to scar formation or hypertrophic scars.
* Those who have joined other clinical trials such ass medical device related and other similar trials within the past six months.
* Those with a medical history of cosmetic filling agent allergy, any type of hyaluronic acid implants, or drugs (such as antibiotics, antihistamine, non-steroidal anti-inflammatory analgesics), or those with a medical history of local anesthetic allergy.
* Patients undergoing anticoagulant treatment, those who have a medical history of coagulation defects, or those taking Chinese medicine for promoting blood circulation.
* Those whose medication and medical conditions are deemed unfit for inclusion in the research based on the judgment of the researcher.
* Those who are unable to comply with re-visit schedule or are unwell to sign the informed consent.

Ages: 30 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 98 (Actual)
Dates: Start 2014-02-13 (Actual); Primary Completion 2015-03-15 (Actual); Study Completion 2015-06-30 (Actual)

PRIMARY OUTCOMES:
WSRS improvement ratio at week 24 post-injection | Baseline and week 24
  The difference of WSRS(Wrinkle Severity Rating Scales) between baseline and week 24. A positive value indicated "effective" improvement; while a value of 0 or a negative value was regarded as "ineffective" treatment. And the WSRS improvement ratio was defined as the effective improvement ratio of either group.

SECONDARY OUTCOMES:
Difference of WSRS score | Baseline to week 24 post-injection
  Based on the photographs, blinded physician rated the score of WSRS (Wrinkle Severity Rating Scales) for both group respectively. The WSRS is a 5-grade instrument for facial wrinkle, Grade 1(absent, no visible nasolabial fold; continuous skin line ) to Grade 5(extreme, extremely deep and long nasolabial fold, detrimental to facial appearance; 2-4mm visible V-shaped fold when stretched; unlikely to have satisfactory correction with injectable implant alone) And the difference of WSRS score was calculated as week 2, 4, 12 and 24 subtracted from baseline.
GAIS score | Baseline to week 24 post-injection
  Compared with the baseline photographs, blinded physician rated the class of GAIS(Global Aesthetic Improvement Scale) from 5(exceptional improvement, excellent corrective result) to 1(worsened patient, the appearance has worsened compared with the original condition) for both group respectively. And the difference of GAIS score was assessed at week 2, 4, 12 and 24.
Difference of Satisfaction of treatment | Baseline to week 24 post-injection
  Subjects rated the points of satisfaction after treatment subjectively from 1(extremely dissatisfied) to 5(extremely satisfied). And the difference of satisfaction was calculated as week 2, 4, 12 and 24 subtracted from baseline.
Incidence of Treatment-related Adverse Events | week 0 to week 52
  The adverse events are defined as any unfavorable sign occurrence in a subject after treatment. The investigator assesses the severity and the relationship of each event to the use of the study device.